CLINICAL TRIAL: NCT07364214
Title: A Phase 1, Open-Label Study to Characterize the Metabolism, Excretion, and Mass Balance of a Single Intravenous Dose of 100 mg Containing 75 µCi of [14C]-Quemliclustat in Healthy Adult Male Participants
Brief Title: Metabolism, Excretion, and Mass Balance Study of Quemliclustat in Healthy Adult Participants (ARC-24)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ARC-24
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: AB680; Quemliclustat; Pharmacokinetics
MeSH Terms: interventions — quemliclustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Quemliclustat (Experimental): Participants will receive a single dose of [14C]-quemliclustat through IV infusion.
  Interventions: Drug: Quemliclustat

INTERVENTIONS:
Drug: Quemliclustat — Administered as specified in the treatment arm

SUMMARY:
The purpose of the study is to investigate the routes of elimination and overall mass balance of 100 mg quemliclustat containing 75 μCi [14C] following a single IV infusion of [14C]-quemliclustat in healthy adult male participants, and to quantify total radioactivity (TRA) in plasma, whole blood, urine, and feces.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, standard vital signs, and ECGs, as deemed by the PI or designee.
* Participants must follow protocol-specified contraception guidance.
* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the start of infusion based on participant self-reporting.
* BMI ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
* Understands the study procedures in the Informed Consent Form and is willing and able to comply with the protocol.

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical, surgical, or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
* History or presence of alcohol or drug abuse within the past 2 years prior to the start of infusion.
* History of presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of total radioactivity excreted in urine and feces | Up to 40 days
Total radioactivity in blood | Up to 40 days
Total radioactivity in plasma | Up to 40 days
Excretion of total radioactivity in urine | Up to 40 days
Excretion of total radioactivity in feces | Up to 40 days

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 54 days
Area Under the Curve From 0 to Last Observed Non-zero Concentration (AUC [0-Last]) for quemliclustat | Up to 40 days
Area Under the Curve From Time '0' Extrapolated to Infinity (AUC[0-inf]) for quemliclustat | Up to 40 days
Maximum Observed Plasma Concentration (Cmax) for quemliclustat | Up to 40 days
Elimination Half-life (t1/2) for quemliclustat | Up to 40 days
Excretion of quemliclustat in urine | Up to 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy